CLINICAL TRIAL: NCT07173101
Title: A Phase II, Double-blind, Randomized, Cross-over Clinical Investigation of the Effects of Semiconductor Embedded Therapeutic Garments on Cancer-related Cognitive Impairment in Breast and Gynecological Cancer Patients
Brief Title: Clinical Investigation of the Effects of Semiconductor Embedded Therapeutic Garments on Cancer-related Cognitive Impairment in Breast and Gynecological Cancer Patients
Acronym: HEADBAND
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: INCREDIWEAR HOLDINGS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCI189692
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Gynecologic Cancer; Cancer-related Cognitive Difficulties
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will blind the participant, the investigator, and the study team to the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semiconductor embedded therapeutic headband (Experimental)
  Interventions: Device: Semiconductor embedded headband
- Sham Headband (Placebo Comparator)
  Interventions: Device: Sham Headband

INTERVENTIONS:
Device: Semiconductor embedded headband — Week 1-3: Participants will be provided with either an active semi-conductor headbands OR a sham headband, absent of semi-conducting fabric. Participants will be instructed to wear them >18 hours per day and report their daily device usage.
  Week 4-5: Washout. Participants will not wear any headbands that were provided.
  Week 6-8: Participants who wore sham headbands in intervention A will be provided with active semi-conductor embedded headbands and instructed to wear them >18 hours per day, and vice versa.
  Arms: Semiconductor embedded therapeutic headband
Device: Sham Headband — Week 1-3: Participants will be provided with either an active semi-conductor headbands OR a sham headband, absent of semi-conducting fabric. Participants will be instructed to wear them >18 hours per day and report their daily device usage.
  Week 4-5: Washout. Participants will not wear any headbands that were provided.
  Week 6-8: Participants who wore sham headbands in intervention A will be provided with active semi-conductor embedded headbands and instructed to wear them >18 hours per day, and vice versa.
  Arms: Sham Headband

SUMMARY:
The purpose of this study is to assess the feasibility of a wearing semiconductor embedded headband for cancer-related cognitive impairment in patients with breast or gynecological cancers. The study will also test the safety and effectiveness of using a semiconductor embedded headband by using a cross-over study design.

The study will consist of the following phases:

* Phase 1: Participants will be randomly assigned to either receive a headband with an active semiconductor or they will receive a sham headband with no semiconductor. They will wear the assigned headband for 18 hours a day for 3 weeks.
* Washout Period: After the first 3-week phase, there will be a 2-week "washout" period. During this time, participants will not wear either headband to allow time for the potential treatment effects to clear from their body.
* Phase 2: After the washout period, participants will switch to the other headband they were previously not receiving. They will wear this assigned headband for 18 hours a day for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 18 years or older.
* Diagnosis of breast or gynecologic cancer.
* Participant has completed chemotherapy within 90 days of enrollment and no additional chemotherapy is planned for the duration of study treatment.
* Perceived cognitive impairment (PCI) score of < 63 in the FACT-Cog-PCI assessment.
* Ability to wear device for at least 18 hours per day during the 6 weeks of intervention.
* ECOG Performance Status ≤ 3.
* Able to speak and understand English.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* History of neurodegenerative conditions, including but not limited to multiple sclerosis, dementia, Alzheimer's, or Parkinson's disease.
* History of CNS diseases such as stroke, meningitis, or traumatic brain injury within 12 months of enrollment.
* Poorly controlled psychological disorders including alcohol dependence, major depressive disorder, schizophrenia, or bipolar disorder.
* Use of tobacco or nicotine products within 90 days of enrollment.
* The diagnosis of another malignancy ≤ 12 months before study enrollment, except for those considered to be adequately treated with no evidence of disease or symptoms and/or will not require therapy during the study duration per treating investigator (i.e., basal cell or squamous cell skin cancer).
* Known brain metastases or cranial epidural disease.
* History of poorly controlled diabetes in the opinion of the investigator.
* Any other condition that would, in the Investigator's judgment, contraindicate the participant's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Active infection requiring systemic therapy.
* Participants taking prohibited medications as described in Section 6.5.1. Cautionary medications may be used as described in Section 6.5.2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of patients that wear the study device for an average of at least 18 hours a day during the study period. For the device to be feasible, this proportion must be at least 75%. | 8 weeks
  The primary objective is to assess the feasibility of wearing semiconductor embedded headbands for cancer-related cognitive impairment in breast and gynecological patients.

SECONDARY OUTCOMES:
The frequency of solicited adverse device effects (ADEs) and unexpected adverse device effects (UADEs) characterized by type. | 8 weeks
  To assess the safety and tolerability of semiconductor embedded headbands in the study population.
The frequency of solicited adverse device effects (ADEs) and unexpected adverse device effects (UADEs) characterized by severity (as defined by the NIH CTCAE, version 5.0). | 8 weeks
  To assess the safety and tolerability of semiconductor embedded headbands in the study population.
The frequency of solicited adverse device effects (ADEs) and unexpected adverse device effects (UADEs) characterized by seriousness. | 8 weeks
  To assess the safety and tolerability of semiconductor embedded headbands in the study population.
The frequency of solicited adverse device effects (ADEs) and unexpected adverse device effects (UADEs) characterized by duration. | 8 weeks
  To assess the safety and tolerability of semiconductor embedded headbands in the study population.
The frequency of solicited adverse device effects (ADEs) and unexpected adverse device effects (UADEs) characterized by relationship to study treatment. | 8 weeks
  To assess the safety and tolerability of semiconductor embedded headbands in the study population.
Change in patient-reported cognitive function as determined by the Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) compared to placebo. | 8 weeks
  To assess the therapeutic effect of semiconductor embedded headbands to reduce cancer-related cognitive impairment (CRCI) symptoms.
Change in processing speed as assessed by the Trail Making Test (TMT). | 8 weeks
  To assess the effect of semiconductor embedded headbands on objective outcome measures in the study population.
Change in executive function as assessed by the Stroop test. | 8 weeks
  To assess the effect of semiconductor embedded headbands on objective outcome measures in the study population.
Change in verbal fluency as assessed by Controlled Oral Word Association Test (COWAT). | 8 weeks
  To assess the effect of semiconductor embedded headbands on objective outcome measures in the study population.
Change in quality of life score as assessed by the EORTC Quality of Life questionnaire. | 8 weeks
  To assess the effect of semiconductor embedded headbands on patient reported outcome measures in the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States